CLINICAL TRIAL: NCT02943863
Title: Comparison of Regional Ventilation Pattern During High Flow Nasal Cannula Between Conventional Low Flow System Nasal Cannula in Patients With Mild to Moderate Hypoxia
Brief Title: Regional Ventilation During High Flow Nasal Cannula and Conventional Nasal Cannula in Patients With Hypoxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Ministry of Trade, Industry & Energy, Republic of Korea (Other Government)
Responsible Party: Principal Investigator, Chae-Man Lim, Professor of Pulmonary and Critical Care Medicine, College of Medicine, University of Ulsan. Chief Director of Intensive Care Units, Asan Medical Center, Asan Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: OMNI
Record Dates: First submitted 2016-10-21; First posted 2016-10-25 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Hypoxia; Oxygen Therapy; High Flow Nasal Cannula; Ventilation
MeSH Terms: conditions — Hypoxia; Respiratory Aspiration

ARMS (2):
- HFNC first (Active Comparator): Patients in "HFNC first" receive oxygen therapy using HFNC in ahead of conventional nasal cannula oxygen therapy. After 20 minutes of HFNC therapy, patients receive conventional nasal cannula oxygen therapy.
  Interventions: Device: HFNC followed by conventional nasal cannula
- LFS first (Active Comparator): Patients in "LFS first" receive oxygen therapy using conventional nasal cannula in ahead of HFNC therapy. After 20 minutes of conventional nasal cannula oxygen therapy, patients receive HFNC oxygen therapy.
  Interventions: Device: Conventional nasal cannula followed by HFNC

INTERVENTIONS:
Device: HFNC followed by conventional nasal cannula
  Arms: HFNC first
Device: Conventional nasal cannula followed by HFNC
  Arms: LFS first

SUMMARY:
High-flow nasal cannula (HFNC) that uses heated and humidified oxygen was recently introduced for bedside care. It has been shown to be associated with reduced risks of tracheal intubation rates and mortality in adult hypoxic patients.

The mechanisms of the effects of HFNC are thought to be related to the favorable effects of the heated and humidified gas, the high-flow rate used to minimize the entrainment of room air, and an increase in the ventilation efficiency, including the elimination of nasopharyngeal dead space, positive end-expiratory pressure (PEEP) effects, and improvements in paradoxical abdominal movement. Regarding the effects on lung volume, global ventilation in the lungs increases during HFNC, which is thought to attribute to PEEP effects. However, how regional ventilation is affected during HFNC in comparison with conventional NC remains unknown.

Because PEEP in mechanically ventilated patients improves the regional homogeneity of ventilation, investigators postulated that HFNC via PEEP effects would result in more homogeneous regional distributions in the ventilation changes. Investigators therefore assessed global and regional ventilation in patients with hypoxia receiving care via HFNC using electric impedance tomography and compared these results with conventional nasal cannula.

ELIGIBILITY:
Inclusion Criteria:

* Age >20 years
* Subjective dyspnea in room air
* SaO2< 90% in room air
* Oxygen requirement for nasal cannula < 6 L/m

Exclusion Criteria:

* Unstable vital signs

  * SBP <90 mmHg
  * DBP < 60 mmHg
  * Heart rate > 120 bpm
  * Respiratory rate > 30 bpm
  * Persistent dyspnea under oxygen therapy using NC
* Severe hypoxia

  * PaO2/FiO2< 200 mmHg
* Unable to cooperate

  * Delirium
  * Reduced cognitive function

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-09; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Tidal variation | Twenty minutes after each oxygen therapy. (At the end of each oxygen therapy)
  Tidal variation using electric impedance tomography

SECONDARY OUTCOMES:
Oxygen saturation | Twenty minutes after each oxygen therapy. (At the end of each oxygen therapy)
  Oxygen saturation at using pulse oxymeter
Respiration Rate | Twenty minutes after each oxygen therapy. (At the end of each oxygen therapy)
Subjective comfort | Twenty minutes after each oxygen therapy. (At the end of each oxygen therapy)
  Subjective comfort using questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Chae-Man Lim, MD, Principal Investigator — Pulmonary and Critical Care Medicine, Asan Medical Center, College of Medicine, University of Ulsan

REFERENCES:
- [Background] Spoletini G, Alotaibi M, Blasi F, Hill NS. Heated Humidified High-Flow Nasal Oxygen in Adults: Mechanisms of Action and Clinical Implications. Chest. 2015 Jul;148(1):253-261. doi: 10.1378/chest.14-2871. PMID 25742321
- [Background] Riera J, Perez P, Cortes J, Roca O, Masclans JR, Rello J. Effect of high-flow nasal cannula and body position on end-expiratory lung volume: a cohort study using electrical impedance tomography. Respir Care. 2013 Apr;58(4):589-96. doi: 10.4187/respcare.02086. PMID 23050520
- [Background] Hsu CF, Cheng JS, Lin WC, Ko YF, Cheng KS, Lin SH, Chen CW. Electrical impedance tomography monitoring in acute respiratory distress syndrome patients with mechanical ventilation during prolonged positive end-expiratory pressure adjustments. J Formos Med Assoc. 2016 Mar;115(3):195-202. doi: 10.1016/j.jfma.2015.03.001. Epub 2015 Apr 3. PMID 25843526
- [Derived] Lee DH, Kim EY, Seo GJ, Suh HJ, Huh JW, Hong SB, Koh Y, Lim CM. Global and Regional Ventilation during High Flow Nasal Cannula in Patients with Hypoxia. Acute Crit Care. 2018 Feb;33(1):7-15. doi: 10.4266/acc.2017.00507. Epub 2018 Jan 22. PMID 31723854